CLINICAL TRIAL: NCT03667690
Title: A Phase 3, Multicenter, Randomized, Double-blind Study of the Efficacy and Safety of Rezafungin for Injection vs. Intravenous Caspofungin Followed by Oral Fluconazole Step Down in the Treatment of Subjects With Candidemia and/or Invasive Candidiasis
Brief Title: Study of Rezafungin Compared to Caspofungin in Subjects With Candidemia and/or Invasive Candidiasis
Acronym: ReSTORE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cidara Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CD101.IV.3.05
Record Dates: First submitted 2018-08-30; First posted 2018-09-12 (Actual); Results first posted 2023-01-06 (Actual); Last update posted 2023-01-06 (Actual); Status verified 2022-12

CONDITIONS: Candidemia; Mycoses; Fungal Infection; Invasive Candidiases
Keywords: Mycoses; Candidiasis; Candidiasis, Invasive; Candidemia; Fungemia; Sepsis; Invasive Fungal Infections; Systemic Inflammatory Response Syndrome; Pathologic Processes; Fluconazole; Caspofungin; Echinocandins; Antifungal Agents; Anti-infective Agents; 14-alpha Demethylase Inhibitors; Cytochrome P-450 Enzyme Inhibitors; Enzyme Inhibitors; Molecular Mechanisms of Pharmacological Action; Steroid Synthesis Inhibitors; Physiological Effects of Drugs; Cytochrome P-450 CYP2C9 Inhibitors; Cytochrome P-450 CYP2C19 Inhibitors
MeSH Terms: conditions — Candidemia; Mycoses; Candidiasis, Invasive; Candidiasis; Fungemia; Sepsis; Invasive Fungal Infections; Systemic Inflammatory Response Syndrome; Pathologic Processes | interventions — Rezafungin; Injections; Caspofungin; Fluconazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group 1: Rezafungin for Injection (Experimental): Subjects in Rezafungin treatment group will receive a 400 mg loading dose in Week 1, followed by 200 mg once weekly, for a total of 2 to 4 doses.
  Daily intravenous placebo infusions, when not administered Rezafungin and a daily placebo for oral step-down therapy (first eligibility on Day 4 or later as advised by a site's national/regional/local guidelines) administered every day.
  Interventions: Drug: Rezafungin for Injection; Drug: oral placebo
- Group 2: Caspofungin (Active Comparator): Subjects in caspofungin arm will receive a total treatment of ≥14 days beginning with a single caspofungin 70 mg IV loading dose on Day 1 followed by 50 mg IV once daily up to 28 days. After ≥3 days of caspofungin treatment(or the minimum duration of IV therapy advised by the site's national/regional/local guidelines, whichever is greater), subjects may be switched to oral fluconazole if specific parameters are met.
  If the subject qualifies, then oral step-down therapy of fluconazole (6 mg/kg to the nearest 200 mg) is administered. After switch to oral step down before Day 8, subjects in the caspofungin group will receive IV placebo on Day 8 to preserve the study blind.
  Interventions: Drug: Caspofungin; Drug: Fluconazole; Drug: intravenous placebo

INTERVENTIONS:
Drug: Rezafungin for Injection — Intravenous antifungal therapy
  Arms: Group 1: Rezafungin for Injection
Drug: Caspofungin — Intravenous antifungal therapy
  Other Names: Cancidas
  Arms: Group 2: Caspofungin
Drug: Fluconazole — Oral antifungal therapy
  Other Names: generic fluconazole
  Arms: Group 2: Caspofungin
Drug: intravenous placebo — Normal saline
  Other Names: placebo infusion
  Arms: Group 2: Caspofungin
Drug: oral placebo — Microcrystalline cellulose
  Other Names: encapsulated cellulose
  Arms: Group 1: Rezafungin for Injection

SUMMARY:
The purpose of this pivotal study is to determine if intravenous Rezafungin is efficacious and safe in the treatment of candidemia and/or invasive candidiasis when compared to caspofungin (followed by optional oral fluconazole).

DETAILED DESCRIPTION:
A Phase 3, multicenter, prospective, randomized, double-blind, efficacy and safety study of Rezafungin for Injection versus an active comparator regimen of caspofungin followed by optional oral fluconazole step-down therapy in subjects with candidemia and/or invasive candidiasis.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide written informed consent. If the subject is unable to consent for himself/herself, a legally acceptable representative must provide informed consent on his/her behalf.
2. Males or females ≥18 years of age.
3. Established mycological diagnosis of candidemia and/or invasive candidiasis from a sample taken ≤4 days (96 hours) before randomization defined as

   * ≥1 blood culture positive for yeast or Candida OR
   * Positive test for Candida from a Sponsor-approved rapid in vitro diagnostic (IVD) OR
   * Positive gram stain (or other method of direct microscopy) for yeast or positive culture for Candida spp. from a specimen obtained from a normally sterile site.
4. Presence of one or more systemic signs attributable to candidemia or invasive candidiasis appearing from ≤12 hours prior to the qualifying positive culture through time of randomization.
5. Willing to initiate or continue medical treatment to cure infections, including receipt of antibiotics and surgical procedures, if required.
6. Female subjects of childbearing potential (all female subjects between 18 years <2 years post-menopausal unless surgically sterile) must agree to and comply with using one barrier method (e.g., female condom with spermicide) plus one other highly effective method of birth control, or sexual abstinence while participating in this study. Male subjects must be vasectomized, abstain from sexual intercourse, or agree to use barrier contraception, and also agree not to donate sperm while participating in the study and for 90 days thereafter (and at least 120 days from the last dose of study drug).
7. For Candidemia only subjects, drawing of a set of blood cultures within 12 hours prior to randomization in the study. The result of these blood cultures is not required for inclusion in the study.

Exclusion Criteria:

1. Any of the following forms of invasive candidiasis at baseline:

   1. Septic arthritis in a prosthetic joint (septic arthritis in a native joint is allowed)
   2. Osteomyelitis
   3. Endocarditis or myocarditis
   4. Meningitis, endophthalmitis, chorioretinitis, or any central nervous system infection
   5. Chronic disseminated candidiasis
   6. Urinary tract candidiasis due to ascending Candida infection secondary to obstruction or surgical instrumentation of the urinary tract
2. Received systemic treatment with an antifungal agent at approved doses for treatment of candidemia for >48 hours (e.g., >2 doses of a once daily antifungal agent or >4 doses of a twice daily antifungal agent) ≤4 days (96 hours) before randomization

   a. Exception: Receipt of antifungal therapy to which any Candida spp. isolated in culture is not susceptible
3. Alanine aminotransferase or aspartate aminotransferase levels >10-fold the upper limit of normal
4. Severe hepatic impairment in subjects with a history of chronic cirrhosis (Child-Pugh score >9)
5. Presence of an indwelling vascular catheter or device that cannot be removed or an abscess that cannot be drained and is likely to be the source of candidemia or invasive candidiasis
6. Known hypersensitivity to Rezafungin for Injection, caspofungin, any echinocandin, or to any of their excipients
7. Meets National Cancer Institute Common Terminology Criteria for Adverse Events, version 5, criteria for ataxia, tremor, motor neuropathy, or sensory neuropathy of Grade 2 or higher
8. History of severe ataxia, tremor, or neuropathy or a diagnosis of multiple sclerosis or a movement disorder (including Parkinson's Disease or Huntington's Disease)
9. Planned or ongoing therapy at Screening with a known neurotoxic medication
10. Previous participation in this or any previous rezafungin study
11. Current participation in another interventional treatment trial with an investigational agent
12. Recent use of an investigational medicinal product within 28 days of the first dose of study drug or presence of an investigational device at the time of screening.
13. Pregnant or lactating females
14. The Principal Investigator (PI) is of the opinion the subject should not participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 199 (Actual)
Dates: Start 2018-10-07 (Actual); Primary Completion 2021-10-07 (Actual); Study Completion 2021-10-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Taylor Sandison, MD, MPH, Study Director — Cidara Therapeutics Inc.
Locations (132):
- United States (19):
  - University of Alabama, Birmingham, Alabama
  - UC Davis, Sacramento, California
  - Emory University Hospital, Atlanta, Georgia
  - Augusta University, Augusta, Georgia
  - Johns Hopkins, Baltimore, Maryland
  - Henry Ford Health System, Detroit, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic Hospital-Rochester, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Washington University St. Louis, St Louis, Missouri
  - Mecury Street Medical, Butte, Montana
  - University of North Carolina, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - ID Clinical Research, Ltd., Toledo, Ohio
  - University of Pittsburgh Falk Medical Center, Pittsburgh, Pennsylvania
  - Reading Hospital and Medical Center, West Reading, Pennsylvania
  - The University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Baylor Scott and White Medical Center, Temple, Texas
  - Carilion Clinic, Roanoke, Virginia
- Argentina (5):
  - Alexander Fleming Specialized Medical Institute, Buenos Aires
  - Cordoba Private Hospital, Córdoba
  - Allende Sanatorium, Córdoba
  - Mayo Private Sanatorium, Córdoba
  - Italian Hospital of Mendoza, Mendoza
- Australia (5):
  - Westmead Public Hospital, Northmead, New South Wales
  - Monash Health, Clayton, Victoria
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
  - Alfred Health, Melbourne, Victoria
  - Royal Melbourne Hospital (RMH), Parkville, Victoria
- Belgium (5):
  - Brugmann University Hospital Center, Brussels
  - Erasme Hospital, Brussels
  - University Hospital Brussels, Brussels
  - Saint Luc University Hospital, Brussels
  - University Hospitals Leuven, Campus Gasthuisberg, Leuven
- Bulgaria (3):
  - Multiprofile Hospital for Active Treatment Puls, Blagoevgrad
  - University Multiprofile Hospital for Active Treatment and Emergency Medicine N.I. Pirogov EAD, Sofia, Clinic of Purulent-Septic Surgery, Sofia
  - University Multiprofile Hospital for Active Treatment and Emergency Medicine N.I. Pirogov EAD, Sofia
- China (17):
  - The First Affiliated Hospital of Bengbu Medical College, Bengbu, Anhui
  - The Second People's Hospital of Hefei, Hefei, Anhui
  - The Second Hospital of Anhui Medical University, Hefei, Anhui
  - Chongqing People's Hospital, Chongqing, Chongqing Municipality
  - Guangzhou First People's Hospital, Guangzhou, Guangdong
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - Qingyuan People's Hospital, Qingyuan, Guangdong
  - Zhongnan Hospital of Wuhan University, Wuhan, Hubei
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - Nanjing First Hospital, Nanjing, Jiangsu
  - Zibo Central Hospital, Zibo, Shandong
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - Huashan Hospital Affiliated Fudan University, Shanghai
  - Shanghai Pulmonary Hospital, Shanghai
  - Institute of Hematology and Blood Diseases Hospital, Chinese Academy of Medical Sciences, Tianjin
  - General Hospital of Tianjin Medical University, Tianjin
- Colombia (3):
  - CEQUIN Foundation Cardiomet, Armenia
  - De La Costa Clinic Ltd., Barranquilla
  - University IPS - Leon XIII Clinic, Medellín
- France (10):
  - Amiens Picardie University Hospital - South, Amiens
  - Centre Hospitalier Victor Dupouy - Argenteuil, Argenteuil
  - Roger Salengro Hospital, Lille
  - Marseille University Hospital Center - North Hospital, Marseille
  - Hotel Dieu Hospital Nantes University Hospital Center, Nantes
  - Saint-Louis Hospital, Paris
  - Paris University Hospitals Center - Cochin Hospital, Paris
  - University Hospital Center of Poitiers, Poitiers
  - Civil Hospital of Strasbourg, Strasbourg
  - Tours University Hospital Center, Bretonneau Hospital, Tours
- Germany (3):
  - University Hospital Köln, Cologne
  - University Hospital Freiburg, Freiburg im Breisgau
  - Johannes Gutenberg University Medical Center, Mainz
- Greece (5):
  - General Hospital of Athens "Evangelismos", 5th Department of Internal Medicine and Infectious Diseases Unit, Athens
  - General Hospital of Athens "Evangelismos", Athens
  - General Hospital of Athens "Laikon", Infectious Diseases Unit, Athens
  - General Hospital of Athens "Laikon", Athens
  - General Hospital of Thessaloniki Ippokratio, Thessaloniki
- Israel (9):
  - Bnai Zion Medical Center, Haifa
  - Lady Davis Carmel Medical Center, Haifa
  - Rambam Health Care Campus, Haifa
  - Edith Wolfson Medical Center, Holon
  - Hadassah Medical Center, Jerusalem
  - The Baruch Padeh Medical Center, Nazareth
  - Ziv Medical Center, Safed
  - The Tel Aviv Sourasky Medical Center, Tel Aviv
  - Chaim Sheba Medical Center, Tel Litwinsky
- Italy (9):
  - Polyclinic S. Orsola-Malpighi, Dept. of Organ Impairment and Transplants, Bologna
  - ASST Large Metropolitan Hospital Niguarda, Infectious Diseases Department, Milan
  - University Polyclinic Hospital of Modena, Modena
  - University Hospital of Modena, Modena
  - University of Milano-Bicocca - San Gerardo Hospital, Monza
  - University Polyclinic Hospital "Paolo Giaccone" Palermo, Infectious Disease Department, ICU, Palermo
  - University Polyclinic Foundation Agostino Gemelli - IRCCS, Rome
  - Integrated University Health Authority of Trieste, Trieste
  - Integrated University Hospital "Santa Maria della Misericordia" of Udine, Udine
- Singapore (2):
  - National University Hospital, Singapore
  - Tan Tock Seng Hospital, Singapore
- South Korea (6):
  - Wonju Severance Christian Hospital, Wŏnju, Gangwon-do
  - Dong-A University Hospital, Busan
  - Severance Hospital, Yonsei University Health System, Seoul
  - Samsung Medical Center, Seoul
  - Chung-Ang University Hospital, Seoul
  - Ajou University Hospital, Suwon
- Spain (13):
  - University Hospital Germans Trias i Pujol, Badalona
  - University Hospital Cruces, Barakaldo
  - Hospital del Mar, Department of Infectious Diseases, Barcelona
  - University Hospital Vall d'Hebron (HUVH), Barcelona
  - Hospital Clinic of Barcelona, Barcelona
  - Parc Tauli Health Corporation, Barcelona
  - General University Hospital Gregorio Maranon, Madrid
  - University Hospital Ramon y Cajal, Madrid
  - University Hospital Clinical San Carlos, Madrid
  - La Paz University Hospital, Madrid
  - University Hospital Puerta de Hierro Majadahonda, Majadahonda
  - University Hospital Virgen Macarena, Seville
  - University and Polytechnic Hospital La Fe, Valencia
- Taiwan (5):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - China Medical University Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Linkou Chang Gung Memorial Hospital, Taoyuan
- Thailand (8):
  - King Chulalongkorn Memorial Hospital, Bangkok
  - Rajavithi Hospital, Bangkok
  - Ramathibodi Hospital, Bangkok
  - Siriraj Hospital, Bangkok
  - Maharaj Nakorn Chiang Mai Hospital, Chiang Mai
  - Srinagarind Hospital, Khon Kaen
  - Thammasat University Hospital, Pathum Thani
  - Songklanagarind Hospital, Songkhla
- Turkey (Türkiye) (5):
  - Hacettepe University School of Medicine, Ankara
  - Ankara University School of Medicine, Ankara
  - Istanbul University School of Medicine, Istanbul
  - Marmara University Pendik Training and Research Hospital, Istanbul
  - Medipol Mega University Hospital, Istanbul

REFERENCES:
- [Derived] Huang H, Feng S, Yu Y, Zhang Y, Yuan Y, Cox L, Zhang Y. Efficacy and Safety of Rezafungin Versus Caspofungin for the Treatment of Candidemia and Invasive Candidiasis in a China Cohort of a Double-Blind, Randomised, Phase 3 Trial (ReSTORE China). Mycoses. 2025 Nov;68(11):e70122. doi: 10.1111/myc.70122. PMID 41194465
- [Derived] Honore PM, Bassetti M, Cornely OA, Dupont H, Fortun J, Kollef MH, Pappas P, Pullman J, Vazquez J, Bielicka I, Dickerson S, Manamley N, Sandison T, Thompson GR. Length of hospital and intensive care unit stay in patients with invasive candidiasis and/or candidemia treated with rezafungin: a pooled analysis of two randomised controlled trials. Crit Care. 2024 Nov 11;28(1):361. doi: 10.1186/s13054-024-05152-2. PMID 39529079
- [Derived] Honore PM, Girardis M, Kollef M, Cornely OA, Thompson GR 3rd, Bassetti M, Soriano A, Huang H, Vazquez J, Kullberg BJ, Pappas PG, Manamley N, Sandison T, Pullman J, Nseir S. Rezafungin versus caspofungin for patients with candidaemia or invasive candidiasis in the intensive care unit: pooled analyses of the ReSTORE and STRIVE randomised trials. Crit Care. 2024 Oct 28;28(1):348. doi: 10.1186/s13054-024-05117-5. PMID 39468640
- [Derived] Clarke F, Grenfell A, Chao S, Richards H, Korman T, Rogers B. Use of echinocandin outpatient parenteral antimicrobial therapy for the treatment of infection caused by Candida spp.: utilization, outcomes and impact of a change to weekly dosing. J Antimicrob Chemother. 2024 Nov 4;79(11):2896-2900. doi: 10.1093/jac/dkae302. PMID 39259571
- [Derived] Soriano A, Honore PM, Cornely OA, Chayakulkeeree M, Bassetti M, Haihui H, Dupont H, Kim YK, Kollef M, Kullberg BJ, Manamley N, Pappas P, Pullman J, Sandison T, Dignani C, Vazquez JA, Thompson GR 3rd. Treatment Outcomes Among Patients With a Positive Candida Culture Close to Randomization Receiving Rezafungin or Caspofungin in the ReSTORE Study. Clin Infect Dis. 2024 Sep 26;79(3):672-681. doi: 10.1093/cid/ciae363. PMID 38985561
- [Derived] Smith HL, Bensman TJ, Mishra S, Li X, Dixon CA, Sheikh J, McMaster OG, Joshi A, Rubin DB, Goodwin A, Miller TJ, Danielsen ZY, Syed I, Shukla SJ, Iarikov D, Kim PW, Farley JJ. Regulatory Considerations in the Approval of Rezafungin (Rezzayo) for the Treatment of Candidemia and Invasive Candidiasis in Adults. J Infect Dis. 2024 Aug 16;230(2):505-513. doi: 10.1093/infdis/jiae146. PMID 38502709
- [Derived] Thompson GR 3rd, Soriano A, Honore PM, Bassetti M, Cornely OA, Kollef M, Kullberg BJ, Pullman J, Hites M, Fortun J, Horcajada JP, Kotanidou A, Das AF, Sandison T, Aram JA, Vazquez JA, Pappas PG. Efficacy and safety of rezafungin and caspofungin in candidaemia and invasive candidiasis: pooled data from two prospective randomised controlled trials. Lancet Infect Dis. 2024 Mar;24(3):319-328. doi: 10.1016/S1473-3099(23)00551-0. Epub 2023 Nov 23. PMID 38008099
- [Derived] Thompson GR 3rd, Soriano A, Cornely OA, Kullberg BJ, Kollef M, Vazquez J, Honore PM, Bassetti M, Pullman J, Chayakulkeeree M, Poromanski I, Dignani C, Das AF, Sandison T, Pappas PG; ReSTORE trial investigators. Rezafungin versus caspofungin for treatment of candidaemia and invasive candidiasis (ReSTORE): a multicentre, double-blind, double-dummy, randomised phase 3 trial. Lancet. 2023 Jan 7;401(10370):49-59. doi: 10.1016/S0140-6736(22)02324-8. Epub 2022 Nov 25. PMID 36442484
- [Derived] Ham YY, Lewis JS 2nd, Thompson GR 3rd. Rezafungin: a novel antifungal for the treatment of invasive candidiasis. Future Microbiol. 2021 Jan;16(1):27-36. doi: 10.2217/fmb-2020-0217. PMID 33438477

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1: Rezafungin for Injection: Subjects in Rezafungin treatment group will receive a 400 mg loading dose in Week 1, followed by 200 mg once weekly, for a total of 2 to 4 doses.
  Daily intravenous placebo infusions, when not administered Rezafungin and a daily placebo for oral step-down therapy (first eligibility on Day 4 or later as advised by a site's national/regional/local guidelines) administered every day.
  Rezafungin for Injection: Intravenous antifungal therapy
  oral placebo: Microcrystalline cellulose
- Group 2: Caspofungin: Subjects in caspofungin arm will receive a total treatment of ≥14 days beginning with a single caspofungin 70 mg IV loading dose on Day 1 followed by 50 mg IV once daily up to 28 days. After ≥3 days of caspofungin treatment(or the minimum duration of IV therapy advised by the site's national/regional/local guidelines, whichever is greater), subjects may be switched to oral fluconazole if specific parameters are met.
  If the subject qualifies, then oral step-down therapy of fluconazole (6 mg/kg to the nearest 200 mg) is administered. After switch to oral step down before Day 8, subjects in the caspofungin group will receive IV placebo on Day 8 to preserve the study blind.
  Caspofungin: Intravenous antifungal therapy
  Fluconazole: Oral antifungal therapy
  intravenous placebo: Normal saline
Period: Overall Study
Arm/Group | Group 1: Rezafungin for Injection | Group 2: Caspofungin
Started (Subjects were randomly assigned (1:1 ratio) to receive either rezafungin for injection or caspofungin. Randomization was stratified based on diagnosis (candidemia only; invasive candidiasis) and by Acute Physiology and Chronic Health Evaluation (APACHE II) score/absolute neutrophil count (ANC) (APACHE II score ≥20 OR ANC <500 cells/microliter; APACHE II score <20 AND ANC ≥500 cells/microliter) at screening.) | 100 | 99
Completed Study Drug Regimen Through Study Day 14 (Discontinuations of study drug prior to Day 14 occurred in 34 and 28 subjects in the rezafungin for injection and caspofungin treatment groups, respectively. The primary reasons for study drug discontinuation prior to Day 14 were death and adverse events. Other reasons for study drug discontinuation prior to Day 14 were singular in nature and did not have a clear pattern for reason or relationship to treatment assignment.) | 66 | 71
Completed | 59 | 59
Not Completed | 41 | 40
Not completed — Adverse Event | 0 | 3
Not completed — Death | 22 | 21
Not completed — Lost to Follow-up | 4 | 5
Not completed — Withdrawal by Subject | 7 | 8
Not completed — Subject could not return for additional investigational product | 1 | 0
Not completed — Subject discharged to hospice care | 2 | 0
Not completed — Withdrawal of consent by subject's legally authorized representative; subject placed in hospice | 1 | 0
Not completed — Study visit missed or conducted over the phone due to Coronavirus disease 2019 (COVID-19) pandemic | 2 | 1
Not completed — Diagnosis of other types of invasive candidiasis | 1 | 1
Not completed — Subject was dropped due to exclusion criterion number 9 | 1 | 0
Not completed — Per Medical Monitor, visits performed over the phone were to be considered as early discontinuation | 0 | 1

BASELINE CHARACTERISTICS:
Population: The Intent-to-Treat (ITT) population analyzed consisted of all subjects randomized to treatment. Subjects were analyzed based on the treatment group to which they were randomized.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: Rezafungin for Injection | Group 2: Caspofungin | Total
Number analyzed (Participants) | 100 | 99 | 199
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 60 | 58 | 118
  >=65 years | 40 | 41 | 81
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.5 (15.80) | 62.0 (14.57) | 60.7 (15.22)
Age, Continuous [Median (Full Range); unit: years] | 59.0 [19 to 89] | 62.0 [20 to 91] | 61.0 [19 to 91]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 43 | 76
  Male | 67 | 56 | 123
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 4 | 11
  Not Hispanic or Latino | 89 | 94 | 183
  Unknown or Not Reported | 4 | 1 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 27 | 31 | 58
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 4 | 9
  White | 61 | 60 | 121
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 6 | 3 | 9
Region of Enrollment [Number; unit: participants]
  Australia | 8 | 5 | 13
  Belgium | 5 | 7 | 12
  Bulgaria | 6 | 4 | 10
  China | 6 | 5 | 11
  Colombia | 1 | 0 | 1
  France | 5 | 1 | 6
  Greece | 6 | 11 | 17
  Israel | 3 | 2 | 5
  Italy | 2 | 3 | 5
  Singapore | 3 | 0 | 3
  South Korea | 6 | 6 | 12
  Spain | 12 | 12 | 24
  Taiwan | 3 | 1 | 4
  Thailand | 8 | 17 | 25
  United States | 26 | 25 | 51
Weight [Mean (Standard Deviation); unit: kilograms] — Population: Data was not captured for all subjects, as some subjects did not have weight determined at Screening.
  kilograms
    number analyzed (Participants) | 95 | 91 | 186
    (all) | 73.52 (23.250) | 69.82 (22.602) | 71.71 (22.948)
Weight [Median (Full Range); unit: kilograms] — Population: Data was not captured for all subjects, as some subjects did not have weight determined at Screening.
  kilograms
    number analyzed (Participants) | 95 | 91 | 186
    (all) | 68.00 [37.2 to 149.9] | 66.20 [33.0 to 153.6] | 67.90 [33.0 to 153.6]
Height [Mean (Standard Deviation); unit: centimeters] — Population: Data was not captured for all subjects, as some subjects did not have height determined at Screening.
  centimeters
    number analyzed (Participants) | 94 | 90 | 184
    (all) | 169.51 (9.984) | 167.29 (11.397) | 168.42 (10.727)
Height [Median (Full Range); unit: centimeters] — Population: Data was not captured for all subjects, as some subjects did not have height determined at Screening.
  centimeters
    number analyzed (Participants) | 94 | 90 | 184
    (all) | 170.00 [137.0 to 190.0] | 168.00 [115.0 to 192.0] | 168.00 [115.0 to 192.0]
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilograms/meter^2] — Population: Data was not captured for all subjects, as some subjects did not have BMI calculated at Screening.
  kilograms/meter^2
    number analyzed (Participants) | 94 | 88 | 182
    (all) | 25.43 (7.037) | 24.47 (6.460) | 24.97 (6.763)
Body Mass Index (BMI) [Median (Full Range); unit: kilograms/meter^2] — Population: Data was not captured for all subjects, as some subjects did not have BMI calculated at Screening.
  kilograms/meter^2
    number analyzed (Participants) | 94 | 88 | 182
    (all) | 23.63 [13.7 to 51.9] | 24.07 [12.9 to 47.6] | 24.02 [12.9 to 51.9]
Diagnosis [Count of Participants; unit: Participants]
  Candidemia only | 70 | 68 | 138
  Invasive candidiasis | 30 | 31 | 61
Modified Acute Physiology and Chronic Health Evaluation (APACHE) II Score Category [Count of Participants; unit: Participants] — The APACHE II score is a validated predictor of mortality in critically ill patients. It can be used in clinical trials at baseline to estimate the overall severity of illness in a patient population. Knaus WA, et al. APACHE II: a severity of disease classification system. Crit Care Med. 1985 13(10):818-29. APACHE II score = acute physiology score + age points + chronic health points. Minimum score = 0; maximum score = 71. Subjects were stratified by estimated mortality (as a percentage) based on APACHE II scores: 0-9 (4-8%), 10-19 (15-24%), ≥20 (≥40%).
  Participants
    ≥20 | 15 | 18 | 33
    10-19 | 43 | 44 | 87
    0-9 | 41 | 37 | 78
    Missing | 1 | 0 | 1
Modified Acute Physiology and Chronic Health Evaluation (APACHE) II Score [Mean (Standard Deviation); unit: units on a scale] — The APACHE II score is a validated predictor of mortality in critically ill patients. Knaus WA, et al. APACHE II: a severity of disease classification system. Crit Care Med. 1985 13(10):818-29.APACHE II score = acute physiology score + age points + chronic health points. Minimum score = 0; maximum score = 71. A mean APACHE II score of 0-19 indicates an estimated mortality (as a percentage) of 4-24%, whereas a score ≥20 reflects a more severely ill patient population with estimated mortality ≥40%. Population: Data was not captured for all subjects, as some subjects did not have the modified APACHE II calculation performed.
  units on a scale
    number analyzed (Participants) | 99 | 99 | 198
    (all) | 12.5 (8.01) | 13.1 (7.11) | 12.8 (7.56)
Modified Acute Physiology and Chronic Health Evaluation (APACHE) II Score [Median (Full Range); unit: units on a scale] — The APACHE II score is a validated predictor of mortality in critically ill patients. Knaus WA, et al. APACHE II: a severity of disease classification system. Crit Care Med. 1985 13(10):818-29. APACHE II score = acute physiology score + age points + chronic health points. Minimum score = 0; maximum score = 71. A median APACHE II score of 0-19 indicates an estimated mortality (as a percentage) of 4-24%, whereas a score ≥20 reflects a more severely ill patient population with estimated mortality ≥40%. Population: Data was not captured for all subjects, as some subjects did not have the modified APACHE II calculation performed.
  units on a scale
    number analyzed (Participants) | 99 | 99 | 198
    (all) | 12.0 [0 to 40] | 12.0 [0 to 37] | 12.0 [0 to 40]
Absolute Neutrophil Count (ANC) (per microliter) at Baseline [Count of Participants; unit: Participants]
  <500/μL | 9 | 6 | 15
  ≥500/μL | 88 | 93 | 181
  Missing | 3 | 0 | 3
Modified APACHE II Score/ANC [Count of Participants; unit: Participants]
  APACHE II score ≥20 or ANC <500/μL | 22 | 21 | 43
  APACHE II score <20 and ANC ≥500/μL | 75 | 78 | 153
  Missing | 3 | 0 | 3
Randomization Strata [Count of Participants; unit: Participants]
  Candidemia only, APACHE II score ≥20 or ANC <500/μL | 19 | 17 | 36
  Candidemia only, APACHE II score <20 and ANC ≥500/μL | 51 | 53 | 104
  Invasive candidiasis, APACHE II score ≥20 or ANC <500/μL | 5 | 5 | 10
  Invasive candidiasis, APACHE II score <20 and ANC ≥500/μL | 25 | 24 | 49
Estimated Creatinine Clearance [Mean (Standard Deviation); unit: milliliters (mL)/minute] — Population: Data was not captured for all subjects, as some subjects did not have the creatinine clearance calculation performed.
  milliliters (mL)/minute
    number analyzed (Participants) | 94 | 88 | 182
    (all) | 93.73 (109.485) | 81.83 (62.328) | 87.98 (89.788)
Estimated Creatinine Clearance [Median (Full Range); unit: milliliters (mL)/minute] — Population: Data was not captured for all subjects, as some subjects did not have the creatinine clearance calculation performed.
  milliliters (mL)/minute
    number analyzed (Participants) | 94 | 88 | 182
    (all) | 78.43 [9.4 to 949.6] | 64.93 [0.4 to 314.0] | 72.01 [0.4 to 949.6]
Child-Pugh Score Category [Count of Participants; unit: Participants] — The Child-Pugh score employs 5 clinical measures of liver disease, each being scored 1 to 3 (least to most severe). The sum of the 5 measures is the total Child-Pugh point score. A total score <7 indicates mild hepatic impairment; a score of 7-9 indicates moderate hepatic impairment; and a score >9 indicates severe hepatic impairment. Calculation of the Child-Pugh score was only required for subjects with a history of chronic cirrhosis. Subjects with no medical history of liver disease were included in the 'No History of Liver Disease/Not Calculated' category regardless of Child-Pugh score.
  Participants
    <7 | 0 | 0 | 0
    7-9 | 2 | 6 | 8
    No History of Liver Disease/Not Calculated | 98 | 93 | 191

OUTCOME MEASURES:

1. Primary Outcome: All-Cause Mortality (US FDA Only)
Description: The number and percentage of subjects in each treatment group who are alive and deceased (or with missing data) in the mITT population.
Time Frame: Day 30 (-2 days)
Population: The modified Intent-to-Treat (mITT) Population includes all subjects who had a documented Candida infection based on central laboratory evaluation of a blood culture or a culture from a normally sterile site obtained ≤4 days (96 hours) before randomization and received ≥1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Rezafungin for Injection | Group 2: Caspofungin
Number analyzed (Participants) | 93 | 94
Participants
  Deceased: Known Deceased (subjects who died on or before Day 30) | 19 | 17
  Deceased: Unknown Survival Status | 3 | 3
  Alive | 71 | 74

2. Primary Outcome: Global Response as Assessed by Data Review Committee (EU European Medicines Agency [EMA] Only)
Description: The number and percentage of subjects in each treatment group who have a global response of cure (clinical cure as assessed by the Investigator, radiological cure [for qualifying invasive candidiasis subjects at baseline], and mycological eradication, as confirmed by the Data Review Committee [DRC]), failure and indeterminate in the mITT population. A global response of cure is indicative of an efficacious outcome and the desired result, whereas a response of failure is indicative of a non-efficacious outcome and the undesired response. Indeterminate responses indicate there was not enough data obtained to determine if the response was cure or failure. Definitions for the global responses of cure, failure, and indeterminate are complex. Detailed definitions for the possible responses to this outcome measure type are provided in Table 7 (Global Response) of the clinical protocol.
Time Frame: Day 14 (±1 day)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Rezafungin for Injection | Group 2: Caspofungin
Number analyzed (Participants) | 93 | 94
Participants
  Cure | 55 | 57
  Failure | 28 | 29
  Indeterminate | 10 | 8

3. Secondary Outcome: Global Response as Assessed by Data Review Committee (US FDA Only)
Description: as for outcome 2
Time Frame: Day 14 (±1 day)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Rezafungin for Injection | Group 2: Caspofungin
Number analyzed (Participants) | 93 | 94
Participants
  Cure | 55 | 57
  Failure | 28 | 29
  Indeterminate | 10 | 8

4. Secondary Outcome: All-Cause Mortality (EU EMA Only)
Description: as for outcome 1
Time Frame: Day 30 (-2 days)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Rezafungin for Injection | Group 2: Caspofungin
Number analyzed (Participants) | 93 | 94
Participants
  Deceased: Known Deceased (subjects who died on or before Day 30) | 19 | 17
  Deceased: Unknown Survival Status | 3 | 3
  Alive | 71 | 74

5. Secondary Outcome: Comparison of Global Response (as Assessed by the DRC) by Visit
Description: as for outcome 2
Time Frame: Day 5, Day 30 (-2 days), End of Treatment (EOT) (≤2 days of last dose) and Follow-up (Days 52-59)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Rezafungin for Injection | Group 2: Caspofungin
Number analyzed (Participants) | 93 | 94
Participants
  Day 5: Cure | 52 | 49
  Day 5: Failure | 32 | 37
  Day 5: Indeterminate | 9 | 8
  Day 30 (-2 days): Cure | 46 | 46
  Day 30 (-2 days): Failure | 31 | 36
  Day 30 (-2 days): Indeterminate | 16 | 12
  EOT (≤2 days of last dose): Cure | 56 | 59
  EOT (≤2 days of last dose): Failure | 29 | 32
  EOT (≤2 days of last dose): Indeterminate | 8 | 3
  Follow-up (Days 52-59): Cure | 42 | 39
  Follow-up (Days 52-59): Failure | 38 | 42
  Follow-up (Days 52-59): Indeterminate | 13 | 13

6. Secondary Outcome: Comparison of Mycological Eradication by Visit
Description: The number and percentage of subjects in each treatment group who have a mycological response of eradication, failure, or indeterminate in the mITT population. A mycological response of eradication means clearance of objective evidence of infection and is indicative of an efficacious outcome and the desired result, whereas a response of failure is indicative of a non-efficacious outcome and the undesired response. Indeterminate responses indicate there was not enough data obtained to determine if the response was eradication or failure. Definitions for the mycological responses of eradication, failure, and indeterminate are complex. Detailed definitions for the possible responses to this outcome measure type are provided in Table 8 (Mycological Response) of the clinical protocol.
  Note: Eradication includes both documented and presumed eradication.
Time Frame: Day 5, Day 14 (±1 day), Day 30 (-2 days), End of Treatment (EOT) (≤2 days of last dose), and Follow-up (Days 52-59)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Rezafungin for Injection | Group 2: Caspofungin
Number analyzed (Participants) | 93 | 94
Participants
  Day 5: Eradication | 64 | 58
  Day 5: Failure | 25 | 27
  Day 5: Indeterminate | 4 | 9
  Day 14 (±1 day): Eradication | 63 | 62
  Day 14 (±1 day): Failure | 26 | 28
  Day 14 (±1 day): Indeterminate | 4 | 4
  Day 30 (-2 days): Eradication | 56 | 53
  Day 30 (-2 days): Failure | 33 | 38
  Day 30 (-2 days): Indeterminate | 4 | 3
  EOT (≤2 days of last dose): Eradication | 63 | 63
  EOT (≤2 days of last dose): Failure | 26 | 29
  EOT (≤2 days of last dose): Indeterminate | 4 | 2
  Follow-up (Days 52-59): Eradication | 48 | 49
  Follow-up (Days 52-59): Failure | 41 | 43
  Follow-up (Days 52-59): Indeterminate | 4 | 2

7. Secondary Outcome: Comparison of Investigators' Assessment of Clinical Response by Visit
Description: The number and percentage of subjects in each treatment group for whom the Investigator determined a clinical response of cure, failure, or indeterminate in the mITT population. A clinical response of cure, as assessed by the Investigator, is indicative of an efficacious outcome and the desired result, whereas a response of failure is indicative of a non-efficacious outcome and the undesired response. Indeterminate responses indicate there was not enough data obtained to determine if the response was cure or failure. Definitions for the clinical responses of cure, failure, and indeterminate are complex. Detailed definitions for the possible responses to this outcome measure type are provided in Table 9 (Investigator's Assessment of Clinical Response) of the clinical protocol.
Time Frame: Day 5, Day 14 (±1 day), Day 30 (-2 days), End of Treatment (EOT) (≤2 days of last dose), and Follow-up (Days 52-59)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Rezafungin for Injection | Group 2: Caspofungin
Number analyzed (Participants) | 93 | 94
Participants
  Day 5: Cure | 59 | 70
  Day 5: Failure | 31 | 22
  Day 5: Indeterminate | 3 | 2
  Day 14 (±1 day): Cure | 62 | 63
  Day 14 (±1 day): Failure | 26 | 27
  Day 14 (±1 day): Indeterminate | 5 | 4
  Day 30 (-2 days): Cure | 51 | 52
  Day 30 (-2 days): Failure | 32 | 34
  Day 30 (-2 days): Indeterminate | 10 | 8
  EOT (≤2 days of last dose): Cure | 65 | 64
  EOT (≤2 days of last dose): Failure | 22 | 26
  EOT (≤2 days of last dose): Indeterminate | 6 | 4
  Follow-up (Days 52-59): Cure | 46 | 44
  Follow-up (Days 52-59): Failure | 38 | 40
  Follow-up (Days 52-59): Indeterminate | 9 | 10

8. Secondary Outcome: Comparison of Radiological Response by Investigator by Visit
Description: The number and percentage of subjects with invasive candidiasis (documented by radiologic/imaging evidence at baseline) in each treatment group who have a radiological response (as assessed by the Investigator) of cure, failure, and indeterminate in the mITT population. A radiological response of cure is indicative of an efficacious outcome and the desired result, whereas a response of failure is indicative of a non-efficacious outcome and the undesired response. Indeterminate responses indicate there was not enough data obtained to determine if the response was cure or failure. Definitions for the radiological responses of cure, failure, and indeterminate are complex. Detailed definitions for the possible responses to this outcome measure type are provided in Table 10 (Radiological Response) of the clinical protocol.
Time Frame: Day 5, Day 14 (±1 day), Day 30 (-2 days), End of Treatment (EOT) (≤2 days of last dose), and Follow-up (Days 52-59)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Rezafungin for Injection | Group 2: Caspofungin
Number analyzed (Participants) | 17 | 17
Participants
  Day 5: number analyzed (Participants) | 15 | 17
  Day 5: Cure | 4 | 6
  Day 5: Failure | 2 | 2
  Day 5: Indeterminate | 9 | 9
  Day 14 (±1 day): Cure | 11 | 10
  Day 14 (±1 day): Failure | 2 | 6
  Day 14 (±1 day): Indeterminate | 4 | 1
  Day 30 (-2 days): Cure | 10 | 11
  Day 30 (-2 days): Failure | 4 | 6
  Day 30 (-2 days): Indeterminate | 3 | 0
  EOT (≤2 days of last dose): number analyzed (Participants) | 16 | 17
  EOT (≤2 days of last dose): Cure | 9 | 11
  EOT (≤2 days of last dose): Failure | 2 | 6
  EOT (≤2 days of last dose): Indeterminate | 5 | 0
  Follow-up (Days 52-59): Cure | 12 | 10
  Follow-up (Days 52-59): Failure | 3 | 7
  Follow-up (Days 52-59): Indeterminate | 2 | 0

9. Secondary Outcome: Number of Subjects With Treatment-Emergent Adverse Events [Safety and Tolerability]
Description: The number and percentage of subjects in each treatment group that experienced at least one treatment-emergent adverse event (TEAE) based on clinical chemistry, hematology and urine analysis laboratory test, vital sign, physical exams and electrocardiogram (ECG) abnormalities.
  Notes: A subject with multiple adverse events (AEs) was counted only once. TEAE was defined as an AE that occurred during or after study drug administration and up through the Follow-up visit. The maximum severity and strongest relationship were counted for subjects with multiple events.
Time Frame: Day 1 through Follow-up Visit (Days 52-59)
Population: The Safety Population includes all subjects who received any amount of the study drug. Safety analyses were performed on the Safety Population. Subjects who received the wrong study drug for their entire course of study drug were analyzed in the treatment group based on the drug received. Subjects who received the wrong study drug for part of their course of study drug were analyzed in the treatment group based on majority of (i.e., most frequent) doses received.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Rezafungin for Injection | Group 2: Caspofungin
Number analyzed (Participants) | 98 | 98
Participants
  At least one TEAE | 89 | 83
  At least one TEAE up through Day 7 | 68 | 61
  At least one study drug-related TEAE | 16 | 9
  At least one grade 4/5 TEAE | 36 | 37
  At least one TEAE leading to interruption of study drug | 3 | 1
  At least one TEAE leading to discontinuation of study drug | 13 | 11
  At least one TEAE leading to study discontinuation | 20 | 17

10. Secondary Outcome: Evaluate Pharmacokinetics (Cmax)
Description: Evaluate the maximum plasma concentration (Cmax) of rezafungin for injection.
Time Frame: Day 1, 10 minutes before the end of infusion
Population: The Pharmacokinetic (PK) Population includes all subjects who received any amount of study drug and had at least one blood sample with measurable concentrations.
  Note: Although blood samples were collected from all subjects receiving study drug, only PK samples from subjects receiving rezafungin for injection were analyzed.
Measure: Mean (Standard Deviation); unit: micrograms/milliliter
Arm/Group | Group 1: Rezafungin for Injection
Number analyzed (Participants) | 86
micrograms/milliliter | 24.18 (32.497)

11. Secondary Outcome: Evaluate Pharmacokinetics (Cmin)
Description: Evaluate the minimum plasma concentration (Cmin) of rezafungin for injection.
Time Frame: Day 8, pre-dose, within 30 minutes prior to the start of infusion
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: micrograms/milliliter
Arm/Group | Group 1: Rezafungin for Injection
Number analyzed (Participants) | 65
micrograms/milliliter | 2.94 (2.656)

12. Secondary Outcome: Evaluate Pharmacokinetics (Cmin)
Description: Evaluate the minimum plasma concentration (Cmin) of rezafungin for injection.
Time Frame: Day 15, pre-dose, within 30 minutes prior to the start of infusion
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: micrograms/milliliter
Arm/Group | Group 1: Rezafungin for Injection
Number analyzed (Participants) | 16
micrograms/milliliter | 2.81 (1.378)

13. Secondary Outcome: Evaluate Pharmacokinetics (Cmin)
Description: Evaluate the minimum plasma concentration (Cmin) of rezafungin for injection.
Time Frame: Day 22, pre-dose, within 30 minutes prior to the start of infusion
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: micrograms/milliliter
Arm/Group | Group 1: Rezafungin for Injection
Number analyzed (Participants) | 5
micrograms/milliliter | 3.74 (1.948)

ADVERSE EVENTS:
Time Frame: Deaths and adverse events (AEs) were monitored and recorded from the time a subject signed the informed consent form (ICF) through the Follow-up visit (Days 52-59). Non-treatment-emergent adverse events were AEs occurring prior to dosing; treatment-emergent adverse events (TEAEs) were AEs that occurred during or at any time after dosing.
Description: All-Cause Mortality, Serious Adverse Events, and Other (Not Including Serious) Adverse Events were assessed in the Safety Population, which included all subjects who received any amount of the study drug. All safety analyses were performed by actual treatment received.
Arm/Group | Group 1: Rezafungin for Injection | Group 2: Caspofungin
All-Cause Mortality (participants affected / at risk) | 29/98 | 25/98
Serious Adverse Events (participants affected / at risk) | 55/98 | 52/98
Other Adverse Events (participants affected / at risk) | 90/98 | 66/98
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1: Rezafungin for Injection (N=98) | Group 2: Caspofungin (N=98)
Cardiac arrest (Cardiac disorders) | 3 | 0
Cardio-respiratory arrest (Cardiac disorders) | 1 | 1
Cardiopulmonary failure (Cardiac disorders) | 1 | 0
Myocarditis (Cardiac disorders) | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 1 | 1
Intestinal ischaemia (Gastrointestinal disorders) | 0 | 1
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 0 | 2
Multiple organ dysfunction syndrome (General disorders) | 5 | 2
Death (General disorders) | 2 | 0 — Incudes 1 serious adverse event described as Death NOS (not otherwise specified)
Septic shock (Infections and infestations) | 8 | 8
Sepsis (Infections and infestations) | 2 | 4
Bronchopulmonary aspergillosis (Infections and infestations) | 1 | 0
Candida sepsis (Infections and infestations) | 1 | 0
Catheter bacteraemia (Infections and infestations) | 1 | 0
Device related sepsis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 4 | 3
Pneumonia pseudomonal (Infections and infestations) | 1 | 0
Acinetobacter sepsis (Infections and infestations) | 0 | 1
Bacterial sepsis (Infections and infestations) | 0 | 2
COVID-19 (Infections and infestations) | 0 | 1
COVID-19 pneumonia (Infections and infestations) | 0 | 2
Klebsiella sepsis (Infections and infestations) | 0 | 3
Pneumonia klebsiella (Infections and infestations) | 0 | 1
Gastric cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma of the tongue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonia lipoid (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 4
Shock (Vascular disorders) | 2 | 0
Bacteraemia (Infections and infestations) | 2 | 1
Abdominal abscess (Infections and infestations) | 1 | 3
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 2
Acute kidney injury (Renal and urinary disorders) | 1 | 3
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 | 0
Splenic haemorrhage (Blood and lymphatic system disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 1 | 0
Left ventricular dysfunction (Cardiac disorders) | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 1
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 1
Colonic fistula (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Diverticulum (Gastrointestinal disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 1 | 0
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 1
Haemoperitoneum (Gastrointestinal disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 1
Large intestine perforation (Gastrointestinal disorders) | 0 | 1
Proctitis (Gastrointestinal disorders) | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Asthenia (General disorders) | 0 | 1
Complication associated with device (General disorders) | 2 | 0
Fatigue (General disorders) | 1 | 0
Hernia (General disorders) | 0 | 1
Hepatic haemorrhage (Hepatobiliary disorders) | 1 | 0
Hepatic infarction (Hepatobiliary disorders) | 0 | 1
Hypertransaminasaemia (Hepatobiliary disorders) | 0 | 1
Liver injury (Hepatobiliary disorders) | 0 | 1
Anaphylactic shock (Immune system disorders) | 0 | 1
Abdominal infection (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 1 | 0
Cryptococcosis (Infections and infestations) | 1 | 0
Endocarditis (Infections and infestations) | 1 | 0
Enterococcal sepsis (Infections and infestations) | 0 | 1
Fusarium infection (Infections and infestations) | 1 | 0
Meningitis (Infections and infestations) | 0 | 1
Peritonitis (Infections and infestations) | 1 | 0
Pseudomonal sepsis (Infections and infestations) | 0 | 1
Pyelonephritis (Infections and infestations) | 0 | 1
Septic pulmonary embolism (Infections and infestations) | 0 | 1
Systemic candida (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Vascular device infection (Infections and infestations) | 0 | 1
Abdominal wound dehiscence (Injury, poisoning and procedural complications) | 1 | 0
Drain site complication (Injury, poisoning and procedural complications) | 0 | 1
Gastrointestinal anastomotic leak (Injury, poisoning and procedural complications) | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 1 | 0
Weight decreased (Investigations) | 0 | 1
Alkalosis hypochloraemic (Metabolism and nutrition disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Hyperglycaemic hyperosmolar nonketotic syndrome (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Haematoma muscle (Musculoskeletal and connective tissue disorders) | 0 | 1
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 1 | 0
Encephalopathy (Nervous system disorders) | 0 | 1
Hypertensive encephalopathy (Nervous system disorders) | 0 | 1
Subarachnoid haemorrhage (Nervous system disorders) | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 1 | 0
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Red man syndrome (Skin and subcutaneous tissue disorders) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0
Circulatory collapse (Vascular disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 0
Hypovolaemic shock (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1: Rezafungin for Injection (N=98) | Group 2: Caspofungin (N=98)
Pyrexia (General disorders) | 14 | 5
Hypokalaemia (Metabolism and nutrition disorders) | 12 | 9
Anaemia (Blood and lymphatic system disorders) | 9 | 9
Hypomagnesaemia (Metabolism and nutrition disorders) | 7 | 3
Diarrhoea (Gastrointestinal disorders) | 6 | 7
Pneumonia (Infections and infestations) | 6 | 1
Vomiting (Gastrointestinal disorders) | 6 | 2
Abdominal pain (Gastrointestinal disorders) | 5 | 4
Constipation (Gastrointestinal disorders) | 5 | 3
Hypophosphataemia (Metabolism and nutrition disorders) | 5 | 4
Nausea (Gastrointestinal disorders) | 5 | 2
Hypotension (Vascular disorders) | 4 | 6
Urinary tract infection (Infections and infestations) | 4 | 6
Acute kidney injury (Renal and urinary disorders) | 2 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2020-10-15): https://cdn.clinicaltrials.gov/large-docs/90/NCT03667690/Prot_000.pdf
  • Statistical Analysis Plan (2021-11-22): https://cdn.clinicaltrials.gov/large-docs/90/NCT03667690/SAP_001.pdf